CLINICAL TRIAL: NCT03678142
Title: DetectAB - Detecting Antibiotics - A Pilot Project
Brief Title: DetectAB - Detecting Antibiotics
Acronym: DetectAB
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-01155; me18Eckstein
Record Dates: First submitted 2018-08-21; First posted 2018-09-19 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Antibiotic Drug Concentration in Sweat
Keywords: antibiotic drug monitoring in sweat
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: analysis of last resort antibiotic drug (Flucloxacillin, Imipenem, Vancomycin or Cefepim) in sweat and blood — blood draw (4.7 ml EDTA) and sweat sample taken (Macroduct Sweat Collecting System)

SUMMARY:
The secretion of different kinds of antibiotic drugs in sweat is investigated. The concentration and pharmacodynamics of antibiotic drugs in sweat and blood will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Ability to understand the purpose of the study, provide signed and dated informed consent and qualify for therapeutic drug monitoring
* In-patients receiving intravenous therapy with last resort antibiotics Cefepim, Floxapen, Imipenem or Vancomycin for at least 24 hours
* Glomerular Filtration Rate >/= 50 ml/Min

Exclusion Criteria:

* Glomerular Filtration Rate < 50 ml/Min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In- patients currently receiving intravenous antibiotic therapy (Cefepim, Flucloxacillin, Imipenem or Vancomycin) at University Hospital Basel/ Switzerland
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change in detection of last resort antibiotic Flucloxacillin in sweat. | sample taken immediately before and 45 minutes after Flucloxacillin application
  detection of Flucloxacillin in sweat by mass spectrometry (proof of concept).
Change in detection of last resort antibiotic Imipenem in sweat. | sample taken immediately before and 60 minutes after Imipenem application
  detection of Imipenem in sweat by mass spectrometry (proof of concept).
Change in detection of last resort antibiotic Vancomycin in sweat. | sample taken immediately before and 5 hours after Vancomycin application
  detection of Vancomycin in sweat by mass spectrometry (proof of concept).
Change in detection of last resort antibiotic Cefepim in sweat. | sample taken immediately before Cefepim application and 2 hours, 4 hours, 6 hours, 8 hours after Cefepim application
  detection of Cefepim in sweat by mass spectrometry (proof of concept).

SECONDARY OUTCOMES:
concentration (yg/ml) of last resort antibiotic Flucloxacillin in sweat. | sample taken immediately before and 45 minutes after Flucloxacillin application
  quantification of Flucloxacillin in sweat by mass spectrometry.
concentration (yg/ml) of last resort antibiotic Imipenem in sweat. | sample taken immediately before and 60 minutes after Imipenem application
  quantification of Imipenem in sweat by mass spectrometry
concentration (yg/ml) of last resort antibiotic Vancomycin in sweat. | sample taken immediately before and 5 hours after Vancomycin application
  quantification of Vancomycin in sweat by mass spectrometry
concentration (yg/ml) of last resort antibiotic Cefepim in sweat. | sample taken immediately before Cefepim application and 2 hours, 4 hours, 6 hours, 8 hours after Cefepim application
  quantification of Cefepim in sweat and blood by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Jens Eckstein, PD Dr. med, Principal Investigator — Chief Clinical Medical Office
Locations (1):
- University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Brasier N, Widmer A, Osthoff M, Mutke M, De Ieso F, Brasier-Lutz P, Wolfe L, Aithal V, Broeckling CD, Prenni J, Eckstein J. Non-invasive Drug Monitoring of beta-Lactam Antibiotics Using Sweat Analysis-A Pilot Study. Front Med (Lausanne). 2020 Aug 25;7:476. doi: 10.3389/fmed.2020.00476. eCollection 2020. PMID 32984371